CLINICAL TRIAL: NCT06301022
Title: Effectiveness and Safety of Finerenone in Chinese CKD Patients Without Diabetes Mellitus: A Real-world Retrospective Study
Brief Title: Effectiveness and Safety of Finerenone in Chinese CKD Patients Without Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: WXZ-Finerenone
Record Dates: First submitted 2024-01-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; finerenone
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background： This study aimed to evaluate the effectiveness and safety of Finerenone in patients with chronic kidney disease (CKD) without diabetes mellitus(DM), however, evidence based on both clinical trails and real-world data are limited.

Methods:

Patients with CKD without DM were enrolled in this study from December 2022 to December 2024. In conjunction with the established treatment regimen for chronic kidney disease (CKD), study participants were additionally administered Finerenone. To evaluate the therapeutic impact and safety profile of the intervention, three primary biomarkers were monitored: 24-hour urinary protein (UTP), estimated glomerular filtration rate (eGFR), and serum potassium (sK+). These parameters were closely measured on a monthly basis, starting from the point of enrollment and continuing for a duration of twelve months or possibly longer.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is a significant global health issue that leads to end-stage renal disease (ESRD) and is associated with rising healthcare costs and high mortality rates. Its prevalence is increasing due to aging populations and the growing rates of diabetes and hypertension. CKD causes severe complications and significantly impairs patients' quality of life. There are notable disparities in CKD incidence and treatment among different socioeconomic groups, and many healthcare systems struggle with the challenges of managing and funding the disease.

In terms of treatment, there is a particular bottleneck in addressing CKD among non-diabetic patients. Currently, the focus for non-diabetic CKD patients is on controlling blood pressure and proteinuria. However, new treatments such as finerenone show promise in reducing CKD progression and cardiovascular risks in diabetic patients. Ongoing research aims to explore the effectiveness of these treatments in non-diabetic CKD patients as well. It is important to note that further studies are required to confirm the safety and efficacy of finerenone in these specific populations.

ELIGIBILITY:
Inclusion Criteria:

* CKD without diabetes

Exclusion Criteria:

* CKD with diabetes

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the medical histories of 43 individuals who received outpatient services at the Department of Nephrology in The First Affiliated Hospital of Harbin Medical University, located in Harbin, China.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
24 hours urinary total protein | before using finerenone, and after using finerenone assessed on a monthly basis, up to 1 year
  24 hours urinary total protein
estimate Gromerular filtration rate | before using finerenone, and after using finerenone assessed on a monthly basis, up to 1 year
  Chinese estimate Gromerular filtration rate
serum potassium | before using finerenone, and after using finerenone assessed on a monthly basis, up to 1 year
  serum potassium level

CONTACTS AND LOCATIONS:
Locations (1):
- First Aaffiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Yes
Types of Data to be Shared:
  1. Individual participant data (IPD) related to treatment allocation, baseline characteristics, monthly 24-hour urinary protein, estimated glomerular filtration rate, and serum potassium level measurements during the 12-month follow-up.
  2. Associated documentation such as the study protocol, statistical analysis plan, and annotated case report forms.
  Data Access Format and Procedures:
  Data will be made available through a secure access system to bonafide researchers upon completion of a formal application process, which includes a review of the proposed research and a signed data access agreement that outlines the terms and conditions of data use.
  Data Availability Time Frame:
  Anonymized IPD will be made available for sharing 18 months after the primary study results have been published to allow sufficient time for the research team to conduct primary analyses.
Supporting Information: Study Protocol
Time Frame: 18 months
Access Criteria: All requests for access to the IPD will be reviewed by the research team to ensure that proposed analyses are scientifically robust, ethical, and capable of contributing meaningful insights to the field.

REFERENCES:
- [Background] Filippatos G, Anker SD, Agarwal R, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Schloemer P, Tornus I, Joseph A, Bakris GL; FIDELIO-DKD Investigators. Finerenone and Cardiovascular Outcomes in Patients With Chronic Kidney Disease and Type 2 Diabetes. Circulation. 2021 Feb 9;143(6):540-552. doi: 10.1161/CIRCULATIONAHA.120.051898. Epub 2020 Nov 16. PMID 33198491

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT06301022/Prot_SAP_000.pdf